CLINICAL TRIAL: NCT06929832
Title: Post-Market Evaluation of Active Thrombectomy and Proximal Aspiration During Lower Extremity Tibial Interventions
Acronym: Protexus 1
Status: Not yet recruiting | Type: Observational
Sponsor: Protexa Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-100
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Post-Market Evaluation of Active Thrombectomy and Proximal Aspiration during Lower Extremity Tibial Interventions

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, open label, single arm post-market clinical study to gather data on the use of the Protexus catheter for temporary blood vessel occlusion while standard of care treatment with other therapeutic devices is conducted in patients undergoing infrapopliteal treatment for peripheral arterial disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject or authorized representative has signed a written Informed Consent
3. Subject is willing to comply with the protocol requirements
4. Rutherford classification 4-6
5. Planned intervention of the native infrapopliteal arteries using balloon angioplasty, atherectomy, and endovascular procedures.
6. Reference vessel diameter for intended location of the distal tip funnel deployment for the Protexus catheter is ≥3.5mm and ≤6.0mm by visual estimate
7. Inflow arteries have ≤30% stenosis. Inflow arteries can be treated at the time of the study procedure to achieve ≤30% stenosis

Exclusion Criteria:

1. Prior intervention within 30 days of treatment in the planned deployment site for the Protexus catheter
2. Presence of a stent in the planned deployment site for the Protexus catheter
3. Has perforation, dissection, or other injury of the access vessel or Protexus catheter deployment site requiring additional stenting or surgical intervention before enrollment
4. History of bleeding diathesis or coagulopathy and unable to receive standard anticoagulation during the index procedure
5. Acute limb ischemia defined as onset of symptoms within two weeks of the planned intervention
6. Inflow arteries have >30% stenosis after treatment at the time of the study procedure
7. Pregnant female subject or subject that has a positive pregnancy test within the previous 7 days
8. Known hypersensitivity or allergy to nitinol
9. Target blood vessels are infected, have extreme tortuosity, or are occluded with calcified material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects being treated for PAD with standard of care interventions
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 30 Days
  The incidence, type, and severity of Protexus related major adverse events (MAEs) through 30-days defined as:
  * Death or organ injury
  * Thrombosis, pseudo-aneurysm, dissection (grade C or greater by visual assessment) or clinical perforation at the Protexus device location
  * Angiographically evident flow limiting distal embolization